CLINICAL TRIAL: NCT00441948
Title: Peterio™ - an Add-on Device for Enhanced Safety of Aesthetic Laser Treatments.
Brief Title: Enhanced Safety Laser Hair Removal System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scilex Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peterio-05
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Hirsutism; Hypertrichosis
Keywords: Hirsutism; Hypertrichosis
MeSH Terms: conditions — Hirsutism; Hypertrichosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Peterio

SUMMARY:
The purpose of this study is to determine whether a new laser system provides better safety and efficacy in hair removal than existing lasers.

DETAILED DESCRIPTION:
Lasers are a well-established, popular modality for removal of unwanted hair. The existing lasers are based on a wavelength that is specifically absorbed by the pigment melanin found in the hair follicle, where the energy is converted to heat resulting in a thermal injury.

However, lasers for hair removal are not without limitations. A laser based long-term hair removal treatment is based on thermal destruction of the hair shaft and follicle using wavelengths that are specifically absorbed by the pigment melanin found in the hair follicle. The heating of hair follicle is done through heat dissipation from the hair shaft. One of the significant limitations of this approach is the fact that the epidermis through which the light energy must penetrate is rich in melanin and therefore absorbs a major portion of the energy, resulting in inadequate heating of the hair follicles. The purpose of the study is an evaluation safety and efficacy of a new laser based device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Fitzpatrick skin types I to VI

Exclusion Criteria:

* Age below 18 or above 75 year old
* Use of photosensitive medications
* Photosensitive diseases
* Active infection of any type and active infection or or a history of Herpes Simplex in the treated site
* Exposure to sun or artificial tanning during the last 3-4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2007-05; Study Completion 2008-04

PRIMARY OUTCOMES:
Hair reduction as counted 1-3 months after each treatment session, depending on the treated area.
Long term clearance will be calculated as the ratio between the value of the baseline hair count taken immediately before the first treatment, and the value obtained at the 3-6 month post treatment hair count.

SECONDARY OUTCOMES:
Measuring treatment discomfort as graded by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Gilad, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Dermatology, Jerusalem, Israel

REFERENCES:
- [Background] Anderson RR, Parrish JA. Selective photothermolysis: precise microsurgery by selective absorption of pulsed radiation. Science. 1983 Apr 29;220(4596):524-7. doi: 10.1126/science.6836297.